CLINICAL TRIAL: NCT02350023
Title: A Randomized Comparative Study of Efficacy and Safety of Topical Latanoprost Versus Topical Corticosteroid in the Treatment of Localized Alopecia Areata
Brief Title: Comparison of Topical Latanoprost vs Topical Corticosteroid in Treatment of Localized Alopecia Areata
Acronym: COLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sonali Bhat, Dr, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9121/PG-2Trg/12/8073
Record Dates: First submitted 2015-01-20; First posted 2015-01-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Alopecia Areata
Keywords: alopecia areata; betamethasone; latanoprost; topical steroid; prostaglandin
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical latanoprost (Active Comparator): Topical latanoprost 0.005%
  Interventions: Drug: Topical latanoprost 0.005%
- Topical betamethasone (Active Comparator): Topical betamethasone 0.05%
  Interventions: Drug: Topical betamethasone 0.05%

INTERVENTIONS:
Drug: Topical latanoprost 0.005% — Local application of the drug on affected skin/scalp
  Arms: Topical latanoprost
Drug: Topical betamethasone 0.05% — Local application of the drug on affected skin/scalp
  Arms: Topical betamethasone

SUMMARY:
Alopecia areata (AA) is an autoimmune disease that involves the hair follicles. Topical corticosteroids are the established agents for treating this disorder. There are several case reports and case series which have demonstrated the efficacy of topical prostaglandins. The two agents have not been compared head-to-head in the published literature. The investigators attempt to compare the efficacy and safety of topical betamethasone and topical latanoprost in the treatment of localised alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an autoimmune disease that involves the hair follicles. Topical corticosteroids are the established agents for treating this disorder. Topical prostaglandins like latanoprost have also been used for this disorder. There are several case reports and case series which have demonstrated the efficacy of topical prostaglandins. However, the two agents i.e. topical corticosteroids and topical latanoprost have not been compared head-to-head in the published literature. The investigators attempt to compare the efficacy and safety of topical betamethasone and topical latanoprost in the treatment of localised alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* • Cases of AA involving scalp and beard area, having 5 or less patches in all, involving less than 40% area

  * Stable disease without appearance of new patch or increase in size of existing patch for at least 15 days

Exclusion Criteria:

* • Pregnant and lactating women

  * Patients on topical treatment for alopecia in the past fifteen days or on systemic treatment for alopecia in the past one month
  * Presence of any contraindication for topical corticosteroids (local skin infections, skin atrophy) or latanoprost (pregnancy, lactation and dermatitis)
  * Any other coexisting hair disorder (viz., trichotillomania, androgenetic alopecia, telogen effluvium)
  * Extensive disease i.e. >5 patches of AA or area involving >40% area / alopecia totalis/ alopecia universalis/ ophiasis

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with hair regrowth (complete, partial, or no regrowth) | 4 months
  Response to the treatment in terms of hair regrowth will be assessed. The reduction in the area affected by alopecia areata will be assessed for each patient

SECONDARY OUTCOMES:
Number of patients suffering from adverse effects | 4 months
  The adverse effects of the study drugs will be assessed including erythema, pruritus, skin atrophy, dermatitis, telangiectasia, and others

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Dermatology, PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Bhat S, Handa S, De D. A randomized comparative study of the efficacy of topical latanoprost versus topical betamethasone diproprionate lotion in the treatment of localized alopecia areata. Indian J Dermatol Venereol Leprol. 2021 Jan-Feb;87(1):42-48. doi: 10.25259/IJDVL_787_19. PMID 33580923